CLINICAL TRIAL: NCT01384864
Title: Endoscopic Multispectral Imaging for the Early Detection of Barrett's Neoplasia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Anandasabapathy, Sharmila, M.D. (Individual)
Collaborators: William Marsh Rice University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GCO# 09-0696 Project 3
Record Dates: First submitted 2011-06-28; First posted 2011-06-29 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Barrett's Esophagus; Intraepithelial Neoplasia
Keywords: barrett's esophagus; intraepithelial neoplasia; cross polarized reflectance examination; vital-dye enhanced fluorescence examination
MeSH Terms: conditions — Barrett Esophagus; Carcinoma in Situ | interventions — Proflavine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment (Experimental): fluorescent imaging with proflavine
  Interventions: Drug: proflavine

INTERVENTIONS:
Drug: proflavine — 2-6 ml of 0.01% proflavine
  Other Names: Proflavine hemisulfate

SUMMARY:
The overall objective of this pilot study is to determine whether multispectral imaging increases the diagnostic accuracy of the current standard of high-definition white-light endoscopy for the detection of Barrett's-associated neoplasia (high grade dysplasia or cancer). The investigators goal is to develop a multispectral endoscopic platform that can be used to survey a large surface area and, potentially, serve as a 'red flag' for microendoscopic imaging of small areas. The goal of this pilot study is to preliminarily determine the accuracy of these modalities during the endoscopic surveillance of Barrett's esophagus.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* known or suspected barrett's esophagus with intraepithelial neoplasia(HGD/cancer)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
to determine whether tissue is neoplastic or non-neoplastic | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States